CLINICAL TRIAL: NCT03736902
Title: Attitudes, Barriers and Facilitators to Physical Activity in People With Multiple Sclerosis Following a Relapse
Brief Title: Views on Physical Activity Following a Relapse in People With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: City, University of London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 248619
Record Dates: First submitted 2018-10-31; First posted 2018-11-09 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: Physical activity; Exercise; Relapse; Exacerbation; Attack
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative semi structured interview — One-to-one semi structured interviews, guided by the Physical Activity for people with a Disability Framework (van der Ploeg et al, 2004) which is a model for understanding the different factors that influence whether people with a disability engage in physical activity. Participants that agree to take part in the study, will be offered an interview either in a private clinic room at the hospital, at their home (if they live within a 40-mile radius of the hospital) or via a web-based video link. The interviews are expected to last one hour and will be conducted by the primary researcher.

SUMMARY:
Multiple Sclerosis (MS) is the most common cause of neurological disability in young adults. Relapsing Remitting Multiple Sclerosis (RRMS) is the most frequent form of MS at the time of diagnosis characterised by relapses, followed by remission. Relapses can result in a sudden change in physical or cognitive symptoms, often impacting a person's ability to function with family, friends and work.

The National Institute for Health and Care Excellence (NICE) Clinical Guidelines for MS recommend encouraging people with MS to exercise regularly but does not provide specific advice on whether exercise should be undertaken during a relapse. Despite the wealth of literature documenting the benefits of exercise for people with MS insufficient evidence exists about exercise during relapse. Research has improved our understanding of what helps people with MS to be physically active and difficulties people encounter but has not provided evidence for how this is affected by a relapse.

The aim of this study is to understand the attitudes of people with MS to physical activity following relapse, including factors that help them to be active and barriers to physical activity. The information gathered will be useful to inform future research and guide the advice health professionals may offer.

Fifteen adults with RRMS who have had a relapse in the preceding 3-4 months will be recruited if their Expanded Disability Status Scale (EDSS) is <7 (EDSS scale is used to quantify disability in MS and monitor changes in the level of disability over time) and they agree to being audio -recorded at interviews. The recruitment will take place at the weekly MS relapse clinic at a hospital in London, UK. Participants will be asked to complete two questionnaires (Patient Determined Disease Steps and the International Physical Activity Questionnaire), answer demographic questions and spend one hour being interviewed by a researcher. It is anticipated the recruitment and interviews be carried out by March 2019.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an inflammatory autoimmune demyelinating disease of the central nervous system (CNS). Over the course of the disease there is usually accompanying axonal degeneration and brain volume loss. It is the most common cause of neurological disability in young adults, with an average age of onset between 20-40 years of age. There are an estimated 107,000 people living with MS in the United Kingdom (UK), with an incidence of 203.4 per 100,000. The aetiology is unknown but is thought to be an interplay between genetic and environmental factors.

MS is an unpredictable condition with varying symptoms depending on the location of damage within the central nervous system. MS is classified into three different phenotypes; relapsing remitting MS (RRMS), secondary progressive MS (SPMS) and primary progressive MS (PPMS). RRMS is the most common form of MS at the time of diagnosis, accounting for 85% of cases. It is characterised by relapses, followed by complete or partial recovery know as a remission. A relapse is defined as 'patient-reported symptoms or objectively observed signs typical of an acute inflammatory demyelinating event in the CNS, current or historical, with duration of at least 24 hours, in the absence of fever or infection'. In people with RRMS, the average relapse frequency is 1.1 per year. Incomplete remissions from a relapse can result in the accumulation of disability. Within 10-15 years 80% of people initially diagnosed with RRMS will transition to SPMS which is characterised by far fewer or no relapses due to less inflammation, but a progressive increase in disability due to neurodegenerative processes. Ten to 15% of people are diagnosed with PPMS, which is defined by a gradual increase in disability from onset, and usually no relapses.

There is no known cure for MS. Disease modifying therapies (DMT's) can alter the immune response which helps control inflammatory activity but their impact on the neurodegenerative processes remains unclear. Steroids are frequently used to treat relapses and consequently the majority of research into relapses has focused on examining their effectiveness and mode of delivery. Steroids can speed up the rate of recovery from a relapse but do not change the level of disability that may occur as a result of the relapse. The majority of improvement in disability following a relapse has been shown to occur within two months but some symptoms, such as arm function, can take up to 12 months.

The most commonly reported symptoms during a relapse are fatigue, lower limb weakness, sensory disturbance and impaired mobility. An MS relapse can result in a sudden change in physical or cognitive symptoms, often impacting on a person's ability to function with family, friends and work. In the UK, a survey of people with MS (PwMS) on their experience of relapses found that 67% of people in paid employment took time off sick and 66% of people required additional support to undertake routine daily tasks following a relapse.

Management of relapses and exacerbations is one of the eight key priorities in the NICE Clinical Guidelines for MS. The guidelines state people having a relapse or exacerbation should be assessed to see if they need additional symptom management or rehabilitation, and whether their care needs have changed. The guidelines also recommend regular exercise but does not provide specific advice on whether exercise should be undertaken during a relapse. In order for PwMS to self-manage effectively whilst they are having a relapse, they need to be given clear information on what they can do to help with their recovery.

Physical activity, which can be defined as 'any bodily movement produced by skeletal muscles that results in energy expenditure', is frequently recommended for PwMS as a way to manage symptoms, improve function, optimise quality of life and reduce the risk of secondary disorders related to inactivity such as heart disease and stroke. Despite physical activity and exercise being promoted as a way to improve symptoms of MS, PwMS typically engage in lower levels of physical activity compared to the general population. Investigating ways to increase activity levels in PwMS is therefore imperative for their long-term health.

There have been a number of studies that have improved our understanding of what helps PwMS to be physically active and what difficulties PwMS encounter. A systematic review of 19 qualitative research studies on physical activity in MS found that the main perceived barriers to being physically active were environmental factors, such as lack of facilities for disabled people and minimal or conflicting advice from health care professionals, and personal barriers, including fatigue and fear. Having a relapse was not cited as barrier. The main facilitators of physical activity have been reported as environmental, including peer support and type of exercise and internal feelings including a sense of accomplishment. Perceived benefits included maintaining physical function, social participation and ability to self-manage. Perceived adverse consequences included increased fatigue and feelings of frustration or inadequacy when exercising. This systematic review gives a clear overview of the barriers, facilitators, benefits and consequences of physical activity in PwMS but does not provide evidence for how this is affected by a relapse which is a point at which PwMS have new or worsening of current symptoms and have expressed feelings of fear and anxiety. In a more recent qualitative study, investigating what PwMS need and want in relation to exercise promotion from healthcare providers, those who were classed as 'sufficiently active' reported wanting advice on how to modify exercise in order to maintain activity levels during a relapse.

Despite the wealth of literature documenting the benefits of exercise for PwMS, there is a paucity of evidence about exercise within the context of relapses. Being physically active has been associated with reduced incidence of relapses, while the occurrence of adverse or serious events associated with exercise for PwMS has been shown to be similar to that of the general adult population. Most research studies involving physical activity or exercise have recent relapse as an exclusion criterion and if participants have a relapse during the study period they are excluded.

There have been two randomised controlled trials evaluating the effectiveness of multidisciplinary therapy (which included exercise) and steroids, compared to steroids alone, which found that multidisciplinary therapy was superior in terms of neurological recovery, functional performance and quality of life. The therapy was individually tailored in these studies which makes it difficult to examine which aspect of the rehabilitation resulted in improvements. Exercise has been shown to be safe outside of the relapse period but little is known about the safety of exercise during a relapse and when physical activity should be reintroduced following a relapse. Consequently, the advice given to people about when to re-engage with physical activity is anecdotal and potentially unclear.

There has been one qualitative study investigating the impact of physical activity on MS symptoms, relapse and disability identity. This study interviewed 15 PwMS to understand the role that physical activity and exercise had on participants daily life, during relapses and the how this was associated with their disability identity. The study did not attempt to investigate the barriers and facilitators to physical activity following a relapse. The results did reveal contradictory findings about the role of exercise in relapses, with some people expressing the belief that exercise could prevent future relapses or that being cardiovascularly fitter would minimise the effect of future relapses, whilst others attributed the cause of their relapse to doing too much exercise. A limitation of this study is that PwMS recruited to the study had previously participated in exercise research, which may have biased the sample towards more physically active participants. Further research is needed into understanding the attitudes of PwMS in the UK to physical activity following a relapse and to explore what helps or hinders them to be physically active following a relapse. This information will help guide advice health professionals may offer and help direct future research into physical activity and exercise following MS relapses.

The proposed study would involve interviewing people with MS who have recently had a relapse to understand more about their attitudes to physical activity and what the barriers and facilitators are to being physically active following a relapse. The participants will be recruited from the MS relapse service at the National Hospital for Neurology and neurosurgery (NHNN) which is part of University College London Hospitals (UCLH). The results from this study will help develop our understanding of physical activity in the context of relapse and will inform future research into physical activity and exercise following MS relapses.

The aim of this research study is to understand the attitudes of PwMS to physical activity following a relapse, including factors that help them to be active and barriers to physical activity.

It is important to learn more about the beliefs and experiences of people engaging in physical activity following a relapse as PwMS report conflicting information from health care professionals. A review of comments on MS internet forums suggests PwMS would like to have more information in relation to physical activity and exercise following a relapse:

'How is one to make sense of the role of exercise during a relapse?' 'When is a return to exercise recommended and for who?' 'How much exercise and what type of exercise [following a relapse]?' 'What can I expect if I exercise [following a relapse]?'

PwMS have also commented that:

'Overdoing exercise can bring on a relapse and will definitely slow down recovery from one.' 'I assumed that anything other than stretching and yoga would prolong recovery.' 'I felt very tired in relapses; exercise would have been very difficult as I needed to save energy for the basic activities of everyday living.' These comments represent conflicting advice on physical activity and exercise following a relapse and demonstrate that PwMS will benefit from clearer advice. However, it is an area with limited evidence to provide people with the answers to their questions. The information obtained from this study will develop our understanding of the attitudes, barriers and facilitators to physical activity following a relapse and will inform the direction that future research into physical activity and exercise following MS relapses should take.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 or over)
* Confirmed diagnosis of Relapsing Remitting Multiple Sclerosis
* Confirmed relapse diagnosed by a consultant neurologist or specialist registrar.
* Relapse within the four months preceding interview date (as most recovery is expected to have occurred by this time)
* Expanded Disability Status Scale (EDSS) score of <7. The EDSS is a 0 - 10 scale used to quantify disability in multiple sclerosis and monitor changes in level of disability over time. A score of 0 represents no disability. The scale is widely used in clinical trials and in the assessment of people with MS. A score of <7 has been chosen as people with a score of ≥7 and above are unable to walk more than five metres and are restricted to a wheelchair for the majority of the daytime and are likely to find it much more difficult to engage in physical activity.
* Agree to be audio-recorded during the interviews
* Patients who speak competent English. This will be assessed initially by the clinical treating team, as patients who can communicate their relapse history in English during the clinic are assumed to have adequate English to participate in this study. In addition, the researcher is an experienced clinical physiotherapist who is exposed to a range of language abilities. If the researcher does not feel the participant has enough English skills to consent, then they will exclude the participant from the study.

Exclusion Criteria:

* Patients who are under the age of 18. Children represent less that 5% of PwMS and their experience is likely to be different to adults.
* Adults unable to participate in an interview spoken in English. Non-English speakers are unable to participate in the study as there are no funds for the hire of interpreters or health advocates, or for the translation of study information or consent documents. In order to gain informed consent, complete the demographic questions, questionnaires and participate in the qualitative interviews with the researcher, participants will need to be able to be able to speak and fluent English.
* People with co-morbidities impacting on physical function in the last year (e.g. heart disease, arthritis, musculoskeletal injury).
* Adults lacking mental capacity to consent to take part in the research.
* People who want to be interviewed at home but live greater than 40 miles radius from the National Hospital for Neurology and Neurosurgery.
* People with a relapse more than four months from the date of interview. This has been chosen so that people that are interviewed have had a recent relapse, with their recovery experience is still fresh in their memory.
* Pseudo-relapse (e.g. from urinary tract infection of lower respiratory tract infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be recruiting from the MS relapse clinic service at a hospital in London, UK. Patients that attend the clinic and meet the inclusion criteria will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Analysis of interview transcripts | 1 year
  Framework analysis (Ritchie and Spencer, 1994)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline McGraw, PhD, Principal Investigator — City, University of London
Locations (1):
- University College London Hospitals, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Mackenzie IS, Morant SV, Bloomfield GA, MacDonald TM, O'Riordan J. Incidence and prevalence of multiple sclerosis in the UK 1990-2010: a descriptive study in the General Practice Research Database. J Neurol Neurosurg Psychiatry. 2014 Jan;85(1):76-84. doi: 10.1136/jnnp-2013-305450. Epub 2013 Sep 19. PMID 24052635
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Vollmer T. The natural history of relapses in multiple sclerosis. J Neurol Sci. 2007 May 15;256 Suppl 1:S5-13. doi: 10.1016/j.jns.2007.01.065. Epub 2007 Mar 7. PMID 17346747
- [Background] Doshi A, Chataway J. Multiple sclerosis, a treatable disease. Clin Med (Lond). 2016 Dec;16(Suppl 6):s53-s59. doi: 10.7861/clinmedicine.16-6-s53. PMID 27956442
- [Background] Motl RW, Sandroff BM, Kwakkel G, Dalgas U, Feinstein A, Heesen C, Feys P, Thompson AJ. Exercise in patients with multiple sclerosis. Lancet Neurol. 2017 Oct;16(10):848-856. doi: 10.1016/S1474-4422(17)30281-8. Epub 2017 Sep 12. PMID 28920890
- [Background] Asano M, Raszewski R, Finlayson M. Rehabilitation interventions for the management of multiple sclerosis relapse: a short scoping review. Int J MS Care. 2014 Summer;16(2):99-104. doi: 10.7224/1537-2073.2013-031. PMID 25061434
- [Background] Perrin Ross A, Williamson A, Smrtka J, Flemming Tracy T, Saunders C, Easterling C, Niewoehner J, Mutschler N. Assessing relapse in multiple sclerosis questionnaire: results of a pilot study. Mult Scler Int. 2013;2013:470476. doi: 10.1155/2013/470476. Epub 2013 May 26. PMID 23766909
- [Background] Hirst CL, Ingram G, Pickersgill TP, Robertson NP. Temporal evolution of remission following multiple sclerosis relapse and predictors of outcome. Mult Scler. 2012 Aug;18(8):1152-8. doi: 10.1177/1352458511433919. Epub 2012 Jan 4. PMID 22217582
- [Background] Nickerson M, Cofield SS, Tyry T, Salter AR, Cutter GR, Marrie RA. Impact of multiple sclerosis relapse: The NARCOMS participant perspective. Mult Scler Relat Disord. 2015 May;4(3):234-40. doi: 10.1016/j.msard.2015.03.005. Epub 2015 Mar 27. PMID 26008940
- [Background] Duddy M, Lee M, Pearson O, Nikfekr E, Chaudhuri A, Percival F, Roberts M, Whitlock C. The UK patient experience of relapse in Multiple Sclerosis treated with first disease modifying therapies. Mult Scler Relat Disord. 2014 Jul;3(4):450-6. doi: 10.1016/j.msard.2014.02.006. Epub 2014 Mar 4. PMID 25877056
- [Background] National Clinical Guideline Centre (UK). Multiple Sclerosis: Management of Multiple Sclerosis in Primary and Secondary Care. London: National Institute for Health and Care Excellence (UK); 2014 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK248064/ PMID 25340249
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Overs S, Hughes CM, Haselkorn JK, Turner AP. Modifiable comorbidities and disability in multiple sclerosis. Curr Neurol Neurosci Rep. 2012 Oct;12(5):610-7. doi: 10.1007/s11910-012-0293-4. PMID 22791240
- [Background] White LJ, Dressendorfer RH. Exercise and multiple sclerosis. Sports Med. 2004;34(15):1077-100. doi: 10.2165/00007256-200434150-00005. PMID 15575796
- [Background] Giovannoni G, Butzkueven H, Dhib-Jalbut S, Hobart J, Kobelt G, Pepper G, Sormani MP, Thalheim C, Traboulsee A, Vollmer T. Brain health: time matters in multiple sclerosis. Mult Scler Relat Disord. 2016 Sep;9 Suppl 1:S5-S48. doi: 10.1016/j.msard.2016.07.003. Epub 2016 Jul 7. PMID 27640924
- [Background] Sandroff BM, Dlugonski D, Weikert M, Suh Y, Balantrapu S, Motl RW. Physical activity and multiple sclerosis: new insights regarding inactivity. Acta Neurol Scand. 2012 Oct;126(4):256-62. doi: 10.1111/j.1600-0404.2011.01634.x. Epub 2012 Jan 3. PMID 22211941
- [Background] Motl RW, McAuley E, Snook EM. Physical activity and multiple sclerosis: a meta-analysis. Mult Scler. 2005 Aug;11(4):459-63. doi: 10.1191/1352458505ms1188oa. PMID 16042230
- [Background] Learmonth YC, Motl RW. Physical activity and exercise training in multiple sclerosis: a review and content analysis of qualitative research identifying perceived determinants and consequences. Disabil Rehabil. 2016;38(13):1227-42. doi: 10.3109/09638288.2015.1077397. Epub 2015 Aug 28. PMID 26314587
- [Background] Wilkinson, H. R. and das Nair, R. (2013), 'The psychological impact of the unpredictability of multiple sclerosis: a qualitative literature meta-synthesis', British Journal of Neuroscience Nursing, 9 (4), pp. 172-178
- [Background] Learmonth YC, Adamson BC, Balto JM, Chiu CY, Molina-Guzman I, Finlayson M, Riskin BJ, Motl RW. Multiple sclerosis patients need and want information on exercise promotion from healthcare providers: a qualitative study. Health Expect. 2017 Aug;20(4):574-583. doi: 10.1111/hex.12482. Epub 2016 Jul 20. PMID 27436592
- [Background] Kjolhede T, Vissing K, Dalgas U. Multiple sclerosis and progressive resistance training: a systematic review. Mult Scler. 2012 Sep;18(9):1215-28. doi: 10.1177/1352458512437418. Epub 2012 Apr 24. PMID 22760230
- [Background] Platta ME, Ensari I, Motl RW, Pilutti LA. Effect of Exercise Training on Fitness in Multiple Sclerosis: A Meta-Analysis. Arch Phys Med Rehabil. 2016 Sep;97(9):1564-1572. doi: 10.1016/j.apmr.2016.01.023. Epub 2016 Feb 16. PMID 26896750
- [Background] Tallner A, Waschbisch A, Wenny I, Schwab S, Hentschke C, Pfeifer K, Maurer M. Multiple sclerosis relapses are not associated with exercise. Mult Scler. 2012 Feb;18(2):232-5. doi: 10.1177/1352458511415143. Epub 2011 Jul 6. PMID 21733890
- [Background] Pilutti LA, Platta ME, Motl RW, Latimer-Cheung AE. The safety of exercise training in multiple sclerosis: a systematic review. J Neurol Sci. 2014 Aug 15;343(1-2):3-7. doi: 10.1016/j.jns.2014.05.016. Epub 2014 May 15. PMID 24880538
- [Background] Bjarnadottir OH, Konradsdottir AD, Reynisdottir K, Olafsson E. Multiple sclerosis and brief moderate exercise. A randomised study. Mult Scler. 2007 Jul;13(6):776-82. doi: 10.1177/1352458506073780. Epub 2007 Mar 15. PMID 17613606
- [Background] Briken S, Gold SM, Patra S, Vettorazzi E, Harbs D, Tallner A, Ketels G, Schulz KH, Heesen C. Effects of exercise on fitness and cognition in progressive MS: a randomized, controlled pilot trial. Mult Scler. 2014 Mar;20(3):382-90. doi: 10.1177/1352458513507358. Epub 2013 Oct 24. PMID 24158978
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Overgaard K, Ingemann-Hansen T. Muscle fiber size increases following resistance training in multiple sclerosis. Mult Scler. 2010 Nov;16(11):1367-76. doi: 10.1177/1352458510377222. Epub 2010 Aug 4. PMID 20685760
- [Background] Craig J, Young CA, Ennis M, Baker G, Boggild M. A randomised controlled trial comparing rehabilitation against standard therapy in multiple sclerosis patients receiving intravenous steroid treatment. J Neurol Neurosurg Psychiatry. 2003 Sep;74(9):1225-30. doi: 10.1136/jnnp.74.9.1225. PMID 12933923
- [Background] Nedeljkovic U, Dackovic J, Tepavcevic DK, Basuroski ID, Mesaros S, Pekmezovic T, Drulovic J. Multidisciplinary rehabilitation and steroids in the management of multiple sclerosis relapses: a randomized controlled trial. Arch Med Sci. 2016 Apr 1;12(2):380-9. doi: 10.5114/aoms.2015.47289. Epub 2015 Mar 18. PMID 27186184
- [Background] Motl RW, Learmonth YC, Pilutti LA, Gappmaier E, Coote S. Top 10 research questions related to physical activity and multiple sclerosis. Res Q Exerc Sport. 2015 Jun;86(2):117-29. doi: 10.1080/02701367.2015.1023099. Epub 2015 Apr 15. PMID 25874730
- [Background] Adamson, B. C., Adamson, M. D., Littlefield, M. M. and Motl, R. W. (2017) 'Move it or lose it: perceptions of the impact of physical activity on multiple sclerosis symptoms, relapse and disability identity', Qualitative Research in Sport, Exercise and Health
- [Background] Overcoming MS (2018) Overcoming MS Forum [Online]. Available at: https://overcomingms.org/forum/viewtopic.php?f=5&t=1214 (Accessed 11 October 2017).
- [Background] Shift MS (2018) Shift MS Forum [Online]. Available at: https://shift.ms/forums/topic/physical-activity-after-a-relapse#post-110842 (Accessed 11 April 2018).
- [Background] MS Society (2017) MS Society Forum [Online]. Available at: https://community.mssociety.org.uk/forums/everyday-living/physical-activity-or-exercise-after-relapse#comment (Accessed 10 April 2018).